CLINICAL TRIAL: NCT02861014
Title: An Open-Label Study To Evaluate the Efficacy and Safety of Ocrelizumab in Patients With Relapsing Multiple Sclerosis Who Have A Suboptimal Response to an Adequate Course of Disease-Modifying Treatment
Brief Title: A Study of Ocrelizumab in Participants With Relapsing Remitting Multiple Sclerosis (RRMS) Who Have Had a Suboptimal Response to an Adequate Course of Disease-Modifying Treatment (DMT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA30005; 2015-005597-38 (EudraCT Number)
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

ARMS (1):
- Ocrelizumab (Experimental): Ocrelizumab will be administered as two 300 mg IV infusions on Days 1 and 15 followed by one 600 mg IV infusions administered at Weeks 24, 48, and 72.
  Interventions: Biological: Ocrelizumab

INTERVENTIONS:
Biological: Ocrelizumab — Ocrelizumab will be administered as two 300 mg IV infusions on Days 1 and 15 followed by one 600 mg IV infusions administered at Weeks 24, 48, and 72.
  Other Names: RO4964913

SUMMARY:
The purpose of this prospective, multicenter, open-label, efficacy, and safety study is to assess the efficacy and safety of ocrelizumab in participants with Relapsing Remitting Multiple Sclerosis (RRMS) who have had a suboptimal response to an adequate course of a Disease-Modifying Treatment (DMT). The study will consist of a Screening period (up to 4 weeks), an Open-label treatment period (96 weeks; with last dose administered at Week 72), and a Follow-up period of at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite diagnosis of RRMS, confirmed as per the revised McDonald 2010 criteria
* Have a length of disease duration, from first symptom, of less than (<) 10 years
* Have received no more than two prior DMTs, and the discontinuation of the most recent DMT was due to lack of efficacy
* Suboptimal disease control while on a DMT
* Expanded Disability Status Scale (EDSS) of 0.0 to 4.0, inclusive, at Screening
* For women of childbearing potential: agreement to use an acceptable birth control method during the treatment period and for at least 6 months after the last dose of study drug

Exclusion Criteria:

* Secondary progressive multiple sclerosis (SPMS) or history of primary progressive or progressive relapsing multiple sclerosis (MS)
* Inability to complete an Magnetic Resonance Imaging (MRI) procedure
* Known presence of other neurological disorders
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History or currently active primary or secondary immunodeficiency
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* History of opportunistic infections
* History or known presence of recurrent or chronic infection
* History of malignancy
* Congestive heart failure
* Known active bacterial, viral, fungal, mycobacterial infection or other infection, excluding fungal infection of nail beds

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 681 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (163):
- St George Hospital, Kogarah, New South Wales, New South Wales, Australia
- Belgium (8):
  - Hospital Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - CHU Tivoli, La Louvière
  - UZ Leuven Gasthuisberg, Leuven
  - Nationaal MS Centrum, Melsbroek
  - Revalidatie en MS Centrum, Overpelt
- Czechia (4):
  - Fakultni nemocnice u sv. Anny; Neurologicka klinika, Brno
  - Nemocnice Jihlava; NEU-Neurologicke oddeleni, Jihlava
  - VFN Praha Poliklinika Rs Centrum - Budova A, Prague
  - Fakultni nemocnice Motol; Neurologicka klinika, Prague
- Denmark (4):
  - Aarhus Universitetshospital, Neurologisk Afd. F, Skleroseklinikken, Aarhus N
  - Rigshospitalet Glostrup; Neurologisk Klinik, Glostrup Municipality
  - Odense Universitetshospital, Neurologisk Afdeling N, Odense C
  - Sydjysk Skleroseklinik - Sønderborg, Sønderborg
- Estonia (3):
  - East Tallinn Central Hospital; Neurology Department, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Finland (2):
  - Terveystalo Tampere, Tampere
  - Mehiläinen Neo Turku, Turku
- France (15):
  - CHU de Besancon Hopital Jean Minjoz; Service de Neurologie, Besançon
  - Groupe Hospitalier Pellegrin; Service de neurochirurgie B, Bordeaux
  - Hopital Neurologique et Neurochirurgical Pierre Wertheimer; Service de Neurologie A, Bron
  - Hopital Gabriel Montpied CHU de Clermont-Ferrand; Service de Neurologie B, Clermont-Ferrand
  - Hopital Roger Salengro; Service de Neurologie, Lille
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - Hôpital Guillaume et René Laënnec; Service Neurologie, Nantes
  - Hôpital Pasteur; Service de Neurologie, Nice
  - Fondation Rothschild; Service de Neurologie, Paris
  - Groupe Hospitalier Pitié- Salpétrière; Service Neurologie, Paris
  - Hôpital Maison Blanche; Service de Neurologie, Reims
  - Hôpitaux Universitaires de strasbourg - hôpital civil, Strasbourg
  - CHU toulouse - Hôpital Purpan; Departement de Neurologie, Toulouse
  - CHRU - Hôpital Bretonneau; Neurologie, Tours
- Germany (38):
  - Klinikum Augsburg, Neurologische Klinik und klinische Neurophysiologie, Augsburg
  - Marianne-Strauß-Klinik; Behandlung Kempfen für Multip Sklero Kranke gemeinnütz GmbH, Berg
  - Charite - Universitatsmedizin Berlin; Klinik fur Neurologie, Berlin
  - Praxis Dr. Said Masri, Berlin
  - Gemeinschaftspraxis Dr.med. Reinhard Ehret/Dr. med Wolfram von Pannwitz, Berlin
  - Jüdisches Krankenhaus Berlin; Abteilung fur Neurologie, Berlin
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Gesundheitszentrum St. Johannes Hospital; Neurolog. Gemeinschaftspraxis Dres. Schmidt, Neudecker etc, Bonn
  - Studienzentrum für Neurologie und Psychiatrie, Böblingen
  - PNP Buchholz, Praxis für Neurologie - Psychiatrie, Dres. Dee/Gößling/Hoge, Buchholz
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Gemeinschaftspraxis für Neurologie; Dr. Katrin Schulte, Dr. Nils Richter, Dr. Margarete Capito, Düsseldorf
  - NeuroCentrum Odenwald; Dres. Reifschneider, Unsorg, Ries, Schumann, Hoffmann, Knoblich, Erbach/Odenwald
  - Universitaetsklinikum Frankfurt; Klinik für Neurologie, Frankfurt
  - Universitätsklinikum Freiburg, Klinik für Neurologie und Neurophysiologie, Freiburg im Breisgau
  - Universiätsklinikum Hamburg-Eppendorf , Multiple Sklerose Tagesklinik u. Ambulanz Neurol. Poliklinik, Hamburg
  - Neurologische Praxisgemeinschaft Hamburger-Straße; Dres. Müller-Habich/Emrich/Vogt, Hamburg
  - MultipEL Studies - Institut für klinische Studien, Hamburg
  - Henriettenstiftung Hannover; Klinik fuer Neurologie und Klinische Neurophysiologie, Hanover
  - Neurologische Klinik, Universitätsklinikum Heidelberg, Heidelberg
  - Oberhavel Kliniken GmbH, Klinik Hennigsdorf, Neurologie, Hennigsdorf
  - Neurozentrum am Klosterforst in Itzehoe, Itzehoe
  - Neurologische Gemeinschaftspraxis Kassel und Vellmar, Ch. Lassek, Dres. Ammerbach, Fetzer, M. Fische, Kassel
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Universitätsklinikum Magdeburg,Otto-von-Guericke-Universität A.ö.R., Klinik für Neurologie, Magdeburg
  - Universitaetsklinikum Mainz - PS; Klinik und Poliklinik fuer Neurologie, Mainz
  - Universitaetsklinikum Marburg; Klinik fuer Neurologie, Marburg
  - Max-Planck-Institut für Psychiatrie, München
  - Klinikum Grosshadern der LMU; Neuroimmunologie II, München
  - Klinikum rechts der Isar der TU Muenchen; Neurologische Klinik und Poliklinik im Neuro-Kopf-Zentrum, München
  - Universitätsklinikum Münster; Klinik und Poliklinik für Neurologie, Münster
  - Ruppiner Kliniken, Hochschulklinikum der Medizinischen Hochschule Brandenburg, Klinik für Neurologie, Neuruppin
  - AMEOS Klinikum Oldenburg, Klinik für Neurologie und Neurophysiologie, Oldenburg in Holstein
  - St. Josefs-Krankenhaus, Klinik für Neurologie, Potsdam
  - NeuroConcept AG C/O mind mvz GmbH, Stuttgart
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
  - NeuroPoint, Gesellschaft für vorbeugende Gesundheitspflege mbH, Ulm
  - Studienzentrum Nordwest, Dr. med. Joachim Springub / Herr Wolfgang Schwarz, Westerstede
- Ireland (3):
  - Cork University Hospital; Clinical Research Facility, Cork
  - Beaumont Hospital, Dublin
  - St Vincents University Hospital, Dublin
- Italy (32):
  - Ospedale SS. Annunziata - Clinica Neurologica - Centro Sclerosi Multipla, Chieti, Abruzzo
  - Ospedale San Salvatore; Clinica Neurologica - Centro Sclerosi Multipla, L’Aquila, Abruzzo
  - Ospedale Dimiccoli Barletta; Dipartimento Testa-Collo - UO Neurologia, Barletta, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; SC Neurologia, San Giovanni Rotondo, Apulia
  - A. O. U. Federico II; Dip Neuroscienze, Scienze Riproduttive ed Odontostomatologiche, Napoli, Campania
  - Università degli Studi della Campania Luigi Vanvitelli; Dip. Ass. Integrato Med Int-II Clinica Neur, Napoli, Campania
  - Ospedale Bellaria; Istituto delle Scienze Neurologiche - UO RIABILITAZIONE SCLEROSI MULTIPLA, Bologna, Emilia-Romagna
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Ospedale S.Camillo Forlanini; UOSD Day Hospital Neurologico e Neurochirurgico, Rome, Lazio
  - Policlinico Universitario A. Gemelli; UOC Neurologia - Centro Sclerosi Multipla, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea; UOC Neurologia, Rome, Lazio
  - Irccs A.O.U.San Martino Ist; Dinogmi, Genoa, Liguria
  - ASST PAPA GIOVANNI XXIII Neurologia USS Malattie Autoimmuni Centro Sclerosi Multipla, Bergamo, Lombardy
  - Ospedale S.Antonio Abate; Neurologia 2 - Sclerosi Multipla e Recupero Neurologico, Gallarate, Lombardy
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico; UOSD Malattie Neurodegenerative, Milan, Lombardy
  - IRCCS Ospedale San Raffaele; Neurologia Neurofisiologia Neuroriabilitazione-Centro Sclerosi Multipla, Milan, Lombardy
  - Fond. Istituto Neurologico C.Besta; UO Neurologia IV - Neuroimmunologia Malattie Neuromuscolari, Milan, Lombardy
  - Ospedale Civile di Montichiari; Centro Sclerosi Multipla, Montichiari, Lombardy
  - IRCCS Istituto Neurologico C. Mondino-Dip. Neurologia Neuroriabilitazione S.S. Sclerosi Multipla, Pavia, Lombardy
  - IRCCS Istituto Neurologico Neuromed; Centro per lo Studio e la Cura della Sclerosi Multipla, Pozzilli, Molise
  - Ospedale Binaghi; Centro Sclerosi Multipla, Cagliari, Sardinia
  - AOU Policlinico V. Emanuele - P.O G. Rodolico; Clinica Neurologica, Centro Sclerosi Multipla, Catania, Sicily
  - Fondazione Istituto S. Raffaele - Giglio; UO Neurologia, Cefalù, Sicily
  - AOU Policlinico Giaccone; UOC Neurologia e Neurofisiopatologia-Amb Sclerosi Multipla, Palermo, Sicily
  - AO Ospedali Riuniti Villa Sofia-Cervello;PO Villa Sofia - UO Neurologia - U.O.S. Neuroimmunologia, Palermo, Sicily
  - AOU Ospedali Riuniti Umberto I-G.M. Lancisi-G. Salesi; SOD Clinica Neurologica-Am.Sclerosi Multipla, Ancona, The Marches
  - AOU Careggi; Neurologia 1-Dip. Neuroscienze Psicologia Area Farmaco Salute del Bambino(NEUROFARBA), Florence, Tuscany
  - AOUC Azienda Ospedaliero-Universitaria Careggi; Neurologia 2, Florence, Tuscany
  - AOU Senese - Presidio Ospedaliero Le Scotte; UOSA Neurologia Sperimentale, Siena, Tuscany
  - AO di Perugia - Ospedale S. Maria della Misericordia; Clinica Neurologica, Perugia, Umbria
  - Azienda Ospedaliera di Padova; Clinica Neurologica, Padua, Veneto
  - Policlinico G.B. Rossi; Dip. Scienze Neurologiche Biomediche - Neurologia B - Amb. Sclerosi Multipla, Verona, Veneto
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Maasstadziekenhuis, Rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - Sint Elizabeth Ziekenhuis, Tilburg
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Sykehuset Buskerud HF; Nevrologisk avdeling, Drammen
- Spain (19):
  - Hospital Universitari de Bellvitge; Servicio de Neurologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General de Castellon; Servicio de Neurología, Castellon, Castellon
  - Hospital Universitari de Girona Dr. Josep Trueta; Servicio de Neurologia, Salt, Girona
  - Complejo Hospitalario Universitario A Coruña (CHUAC); Servicio de Neurologia, A Coruña, LA Coruña
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Neurología, Lleida, Lerida
  - Hospital Quiron de Madrid; Servicio de Neurologia, Pozuelo de Alarcón, Madrid
  - Complejo Hospitalario Universitario de Vigo - Xeral Cies; Servicio de Neurologia, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias; Servicio de Neurología, Oviedo, Principality of Asturias
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Hospital Vall d'Hebron; Servicio de Neurología, Barcelona
  - Hospital Puerta del Mar; Sevicio de Neurologia, Cadiz
  - Universitario de La Princesa; Servicio de Neurología, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Neurología, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Hospital Universitario La Paz; Servicio de Neurologia, Madrid
  - Hospital Universitario Virgen de Arrixaca; Servicio de Neurología, Murcia
  - Hospital Universitario Virgen Macarena; Servicio de Neurologia, Seville
  - Hospital Clinico Universitario de Valencia; Servicio de Neurologia, Valencia
  - Hospital Universitario la Fe; Servicio de Neurologia, Valencia
- Sweden (3):
  - Sahlgrenska Sjukhuset; Neurology, Gothenburg
  - Länssjukhuset Ryhov; Medicinkliniken / Neurologmottagningen, Jönköping
  - Centrum för Neurologi, Stockholm
- Switzerland (2):
  - Universitätsspital Basel Medizin Neurologie; Neurologische Poliklinik, Basel
  - CHUV Lausanne Méd.Neurologie, Lausanne
- Turkey (Türkiye) (8):
  - Hacettepe University Medical Faculty; Neurology, Ankara
  - Istanbul Uni Istanbul Medical Faculty, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi; Noroloji Anabilim Dali, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Hospital; Department of Neurology, Kocaeli
  - Mersin University Medical Faculty; Neurology, Mersin
  - Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun
  - Karadeniz Tecnical Uni. Med. Fac.; Neurology, Trabzon
- United Kingdom (14):
  - New Queen Elizabeth Hospital Birmingham, Birmingham
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Raigmore Hospital, Inverness
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - The Royal London Hospital, London
  - Kings College Hospital, London
  - Charing Cross Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Salford Royal NHS Foundation Trust, Salford
  - Royal Hallamshire Hospita, Sheffield
  - Morriston Hospital, Swansea
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Vermersch P, Oreja-Guevara C, Siva A, Van Wijmeersch B, Wiendl H, Wuerfel J, Buffels R, Kadner K, Kuenzel T, Comi G; CASTING Investigators. Efficacy and safety of ocrelizumab in patients with relapsing-remitting multiple sclerosis with suboptimal response to prior disease-modifying therapies: A primary analysis from the phase 3b CASTING single-arm, open-label trial. Eur J Neurol. 2022 Mar;29(3):790-801. doi: 10.1111/ene.15171. Epub 2021 Nov 25. PMID 34748672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One additional participant was initially enrolled in error and the information provided is based on the ITT population.
Groups:
- Ocrelizumab: Participants received Ocrelizumab as two 300 mg IV infusions on Days 1 and 15 followed by one 600 mg IV infusions administered at Weeks 24, 48, and 72.
Period: Primary Analysis
Arm/Group | Ocrelizumab
Started | 680
Completed | 641
Not Completed | 39
Not completed — Adverse Event | 7
Not completed — Death | 1
Not completed — Lack of Efficacy | 3
Not completed — Physician Decision | 2
Not completed — Pregnancy | 4
Not completed — Protocol Violation | 2
Not completed — Study Terminated By Sponsor | 3
Not completed — Withdrawal by Subject | 14
Not completed — Commercial ocrelizumab | 3
Period: Safety Follow-up
Arm/Group | Ocrelizumab
Started | 64
Completed | 14
Not Completed | 50
Not completed — Adverse Event | 1
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 9
Not completed — Study terminated by sponsor | 1
Not completed — Physician Decision | 1
Not completed — Roll-over to a long term extension study | 1
Not completed — Commercial ocrelizumab | 36

BASELINE CHARACTERISTICS:
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.2 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 436
  Male | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 579
  Unknown or Not Reported | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 625
  More than one race | 2
  Unknown or Not Reported | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With No Evidence of Disease Activity (NEDA) as Per Protocol Defined Events During a 96-Week Period
Description: A protocol-defined event of disease activity was defined by the occurrence of at least one of the following while on treatment with ocrelizumab:
  * A protocol-defined relapse (PDR)
  * 24-week CDP based on increase in EDSS while on treatment with ocrelizumab
  * A T1 Gd-enhanced lesion after Week 8
  * A new and/or enlarging T2 hyperintense lesion on MRI after Week 8 compared to the Week 8 MRI scan
Time Frame: Week 96
Population: The modified intent-to-treat (mITT) population was defined as all participants from the ITT population excluding participants with both screening and the baseline EDSS scores missing.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 658
Percentage of Participants | 74.8 [71.3 to 78.0]

2. Secondary Outcome: Percentage of Participants Free From a Protocol-Defined Event of Disease Activity During 24 Weeks Period
Description: as for outcome 1
Time Frame: Baseline up to 24 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 673
Percentage of Participants | 87.1 [84.3 to 89.5]

3. Secondary Outcome: Percentage of Participants Free From a Protocol-Defined Event of Disease Activity During 48 Weeks Period
Description: as for outcome 1
Time Frame: Baseline up to 48 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 665
Percentage of Participants | 82.6 [79.5 to 85.4]

4. Secondary Outcome: Time to First Protocol-Defined Event of Disease Activity
Description: The definition of a protocol-defined event of disease activity is the occurrence of at least one of the following while on treatment with ocrelizumab:
  * A protocol-defined relapse defined as: Symptoms must persist for >24 hours and should not be attributable to confounding clinical factors; Symptoms should be preceded by neurological stability for at least 30 days; Symptoms should be accompanied by new objective neurological worsening determined with a timely EDSS/ Functional Systems Score (FSS) assessment
  * 24 weeks confirmed disability progression based on increases in EDSS while on treatment with ocrelizumab
  * A T1 Gd-enhanced lesion after Week 8
  * A new and/or enlarging T2 hyperintense lesion on MRI after Week 8 compared to the Week 8 MRI scan.
Time Frame: Baseline up to 96 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Weeks | NA [NA to NA] — Insufficient number of participants with events

5. Secondary Outcome: Change From Baseline to Week 96 in Expanded Disability Status Scale (EDSS)
Description: The EDSS is an ordinal clinical rating scale ranging from 0 (normal neurologic examination) to 10 (death due to MS) in half-point increments.
Time Frame: Baseline, Weeks: 24, 48, 72, 96
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Points on scale
  Baseline | 2.09 (1.06)
  Week 24: number analyzed (Participants) | 679
  Week 24 | -0.02 (0.64)
  Week 48: number analyzed (Participants) | 665
  Week 48 | 0.01 (0.82)
  Week 72: number analyzed (Participants) | 650
  Week 72 | -0.03 (0.85)
  Week 96: number analyzed (Participants) | 640
  Week 96 | -0.01 (0.85)

6. Secondary Outcome: Absolute Change From Baseline in EDSS Category at Week 96
Description: as for outcome 5
Time Frame: Up to Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 640
Percentage of Participants
  Worsened (>0.5) | 13.4
  Stable (Change <= 0.5 and >= -0.5) | 72.2
  Improved (<-0.5) | 14.4

7. Secondary Outcome: Percentage of Participants With a Baseline EDSS Score ≥2 With CDI at Week 96
Description: as for outcome 5
Time Frame: Week 96
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 399
Percentage of Participants | 17.3

8. Secondary Outcome: Annualized Protocol-defined Relapse Rate at Week 96
Time Frame: Week 96
Population: All enrolled participants who received any dose of ocrelizumab were included in the ITT population. Participants who prematurely withdrew from the study for any reason and who did not perform any assessment for any reason were also included in the ITT population.
Measure: Number (95% Confidence Interval); unit: Relapses per participant per year
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Relapses per participant per year | 0.030 [0.023 to 0.038]

9. Secondary Outcome: Time to Onset of 24-week Confirmed Disability Progression
Time Frame: Baseline up to 96 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Weeks | NA [NA to NA] — Insufficient number of participants with events.

10. Secondary Outcome: Time to Onset of First Protocol-Defined Relapse
Description: A protocol-defined multiple sclerosis (MS) relapse is an occurrence of new or worsening neurological symptoms attributable to MS that meets the following criteria:
  * Symptoms must persist for >24 hours and should not be attributable to confounding clinical factors (e.g., fever, infection, injury, adverse reactions to medications)
  * Symptoms should be preceded by neurological stability for at least 30 days
  * Symptoms should be accompanied by new objective neurological worsening determined with a timely EDSS/ Functional Systems Score (FSS) assessment, consistent with an increase of at least:
    * ≥ 0.5 points on EDSS scale
    * or ≥ 2 points on one of the following FSS scales: pyramidal, ambulation, cerebellar, brainstem, sensory, or visual
    * or ≥ 1 point on two or more of the following FSS scales: pyramidal, ambulation, cerebellar, brainstem, sensory, or visual
Time Frame: Baseline up to 96 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Weeks | NA [NA to NA] — Insufficient number of participants with event.

11. Secondary Outcome: Time to Onset of First New and/or Enlarging T2 Lesion
Time Frame: Baseline up to 96 Weeks
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Weeks | NA [NA to NA] — Insufficient number of participants with event.

12. Secondary Outcome: Mean Number of T1 Gd-enhancing Lesions Per MRI Scan at Weeks 24, 48 and 96
Description: Mean number of T1 Gd-enhancing lesions per MRI scan: Total number of T1 Gd-enhanced lesions divided by the total number of interpretable MRI scans
Time Frame: Weeks: 24, 48, 96
Population: All enrolled participants who received any dose of ocrelizumab were included in the ITT population. Participants who prematurely withdrew from the study for any reason and who did not perform any assessment for any reason were also included in the ITT population. Here number of analyzed participants represents participants with data available at given timepoint.
Measure: Mean (95% Confidence Interval); unit: Lesions per scan
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 665
Lesions per scan
  Week 24 | 0.004 [0.001 to 0.014]
  Week 48: number analyzed (Participants) | 658
  Week 48 | 0.004 [0.001 to 0.011]
  Week 96: number analyzed (Participants) | 629
  Week 96 | NA [NA to NA] — No result could be obtained for Week 96, as the model did not converge.

13. Secondary Outcome: Change From Baseline to Week 96 in Total T2 Lesion Volume Detected by Brain MRI From
Time Frame: Baseline, Week 96
Population: All enrolled participants who received any dose of ocrelizumab were included in the ITT population. Participants who prematurely withdrew from the study for any reason and who did not perform any assessment for any reason were also included in the ITT population. Here number of analyzed participants represents participants with data available.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 632
mL | -558.6 (1194.6)

14. Secondary Outcome: Percentage Change From Baseline to Week 96 in Total T2 Lesion Volume Detected by Brain MRI
Time Frame: Baseline, Week 96
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percentage Change From Baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 632
Percentage Change From Baseline | -8.5 (18.2)

15. Secondary Outcome: Volume of New and/or Enlarging T2 Hyperintense Lesions Volume of Lesions Per MRI Scan at Weeks 24, 48, 96
Description: The number of new and/or enlarging T2 lesions at week 24, 48 and 96 is calculated as the sum of the individual number of new and/or enlarging lesions at each visit. Data from other unscheduled assessments is included in this summary or analysis.
Time Frame: Weeks 24, 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: uL
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 670
uL
  Week 24 | 21.4 (241.7)
  Week 48: number analyzed (Participants) | 666
  Week 48 | 23.1 (510.2)
  Week 96: number analyzed (Participants) | 631
  Week 96 | 3.7 (41.6)

16. Secondary Outcome: Mean Number of New and/or Enlarging T2 Hyperintense Lesions Per MRI Scan
Description: Mean number of new and/or enlarging T2 hyperintense lesions per MRI scan: Total number of new and/or enlarging T2 hyperintense lesions divided by the total number of interpretable MRI scans
Time Frame: Weeks 24, 48, 96
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Lesions per scan
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 671
Lesions per scan
  Week 24 | 0.053 [0.038 to 0.075]
  Week 48: number analyzed (Participants) | 666
  Week 48 | 0.009 [0.004 to 0.017]
  Week 96: number analyzed (Participants) | 636
  Week 96 | 0.011 [0.006 to 0.020]

17. Secondary Outcome: Change From Baseline at Week 48 and 96 in T1 Hypointense Lesion Volume
Time Frame: Weeks 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 666
mL
  Week 48 | -416.5 (1224.3)
  Week 96: number analyzed (Participants) | 635
  Week 96 | -528.5 (1144.7)

18. Secondary Outcome: Percentage Change From Baseline at Week 48 and 96 in T1 Hypointense Lesion Volume
Time Frame: Weeks 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 680
Percentage change from baseline
  Week 48: number analyzed (Participants) | 666
  Week 48 | -4.0 (149.7)
  Week 96: number analyzed (Participants) | 635
  Week 96 | -12.5 (21.1)

19. Secondary Outcome: Adjusted Mean Change From Baseline at Week 48 and 96 in T1 Hypointense Lesion Volume
Time Frame: Weeks 48, 96
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 666
mL
  Week 48 | -461.8 [-613.8 to -309.7]
  Week 96: number analyzed (Participants) | 635
  Week 96 | -576.5 [-727.0 to -426.1]

20. Secondary Outcome: Adjusted Mean Percentage Change From Baseline in Brain Volume
Time Frame: Weeks 24, 48, 96
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Mean percentage change from baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 538
Mean percentage change from baseline
  Week 24 | -0.153 [-0.259 to -0.047]
  Week 48: number analyzed (Participants) | 518
  Week 48 | -0.445 [-0.556 to -0.334]
  Week 96: number analyzed (Participants) | 484
  Week 96 | -0.805 [-0.940 to -0.669]

21. Secondary Outcome: Adjusted Mean Percentage Change From Baseline in Cortical Grey Matter Volume
Time Frame: Weeks 48, 96
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Mean percentage change from baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 432
Mean percentage change from baseline
  Week 48 | -0.312 [-0.606 to -0.019]
  Week 96: number analyzed (Participants) | 395
  Week 96 | -0.618 [-0.928 to -0.308]

22. Secondary Outcome: Adjusted Mean Percentage Change From Baseline in White Matter Volume
Time Frame: Weeks 48, 96
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Mean percentage change from baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 432
Mean percentage change from baseline
  Week 48 | -0.382 [-0.609 to -0.154]
  Week 96: number analyzed (Participants) | 395
  Week 96 | -0.745 [-0.983 to -0.507]

23. Secondary Outcome: Mean Change From Baseline in Cognitive Performance (Processing Speed/Working Memory) at Week 48 and Week 96 as Measured by the Brief International Cognitive Assessment for MS - Symbol Digit Modalities Test (SDMT) Score
Description: Brief International Cognitive Assessment for MS (BICAMS) is assessing cognitive processing speed and verbal and visual memory. Symbol Digits Modalities Test (SDMT) is assessing processing speed/working memory. The SDMT presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Participants are asked to voice the digit associated with each symbol as rapidly as possible for 90 sec. There is a single outcome measure - the number correct over the 90 sec time span. The higher the results, the better processing speed/working memory.
Time Frame: Baseline, Weeks: 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Correct responses over 90 seconds
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 610
Correct responses over 90 seconds
  Baseline | 53.8 (13.0)
  Week 48 | 2.5 (9.8)
  Week 96: number analyzed (Participants) | 599
  Week 96 | 1.3 (10.2)

24. Secondary Outcome: Change From Baseline in Cognitive Performance (Visuospatial Memory) at Week 48 and Week 96 as Measured by the Brief International Cognitive Assessment for MS - Brief Visuospatial Memory Test-Revised (BVMT-R) Score
Description: Brief International Cognitive Assessment for MS (BICAMS) is assessing cognitive processing speed and verbal and visual memory. Brief Visuospatial Memory Test-Revised (BVMT-R) is assessing visuospatial memory. In this test, six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. There are three learning trials, and the outcome measure is the total number of points earned over the three learning trials, thus the scale range is 0-36. The higher the result, the better visual/spatial memory.
Time Frame: Baseline, Weeks 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Points on scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 599
Points on scale
  Baseline | 25.0 (6.3)
  Week 48 | -1.9 (5.3)
  Week 96: number analyzed (Participants) | 581
  Week 96 | -1.5 (5.4)

25. Secondary Outcome: Percentage Change From Baseline in Cognitive Performance (Processing Speed/Working Memory) at Week 48 and Week 96 as Measured by the Brief International Cognitive Assessment for MS - Symbol Digit Modalities Test (SDMT) Score
Description: Brief International Cognitive Assessment for MS (BICAMS) is assessing cognitive processing speed and verbal and visual memory. Symbol Digits Modalities Test (SDMT) is assessing processing speed/working memory. The SDMT presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Participants are asked to voice the digit associated with each symbol as rapidly as possible for 90 sec. There is a single outcome measure - the number correct over the 90 sec time span.
Time Frame: Baseline, Weeks 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 610
Percentage change from baseline
  Week 48 | 7.2 (30.8)
  Week 96: number analyzed (Participants) | 599
  Week 96 | 4.8 (30.6)

26. Secondary Outcome: Percentage Change From Baseline in Cognitive Performance (Visuospatial Memory) at Week 48 and Week 96 as Measured by the Brief International Cognitive Assessment for MS - Brief Visuospatial Memory Test-Revised (BVMT-R) Score
Description: as for outcome 24
Time Frame: Baseline, Weeks: 48, 96
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 599
Percentage change from baseline
  Week 48 | -4.4 (31.1)
  Week 96: number analyzed (Participants) | 581
  Week 96 | -2.0 (33.7)

27. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to to 96 weeks after the end of the Treatment Period
Population: Safety analyses were done on the ITT population.
Measure: Number; unit: Percentage of Participants
Groups:
- Ocrelizumab Safety Follow-up: Participants received Ocrelizumab as two 300 mg IV infusions on Days 1 and 15 followed by one 600 mg IV infusions administered at Weeks 24, 48, and 72.
Arm/Group | Ocrelizumab | Ocrelizumab Safety Follow-up
Number analyzed (Participants) | 680 | 64
Percentage of Participants
  Any AE | 89.1 | 57.8
  SAE | 7.2 | 9.4
  Deaths | 0.1 | 0
  AEs leading to study drug discontinuation | 1.0 | NA — During Safety follow-up period participants didn't receive study drug anymore
  SAEs leading to study drug discontinuation | 0.7 | NA — During Safety follow-up period participants didn't receive study drug anymore
  AEs leading to dose modification/interruptionb | 15.0 | NA — During Safety follow-up period participants didn't receive study drug anymore
  Infusion-related reactions (IRRs) | 43.2 | 0
  Serious IRRs | 0.1 | 0
  Infections | 66.9 | 28.1
  Serious infections | 1.6 | 0
  Malignancies | 0.4 | 0
  Pregnancies | 0.7 | 1.5

ADVERSE EVENTS:
Time Frame: From Baseline up to to 96 weeks after the end of the Treatment Period. Time frame includes the safety-follow-up period.
Description: One participant discontinued the study before receiving treatment and was excluded from safety population.
Arm/Group | Ocrelizumab | Ocrelizumab Safety Follow-up
All-Cause Mortality (participants affected / at risk) | 1/680 | 0/64
Serious Adverse Events (participants affected / at risk) | 49/680 | 6/64
Other Adverse Events (participants affected / at risk) | 531/680 | 14/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=680) | Ocrelizumab Safety Follow-up (N=64)
OEDEMA (Gastrointestinal disorders) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (2)
DEPRESSION SUICIDAL (Psychiatric disorders) | 0 (0) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GRANULOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 (1) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CROHN'S DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
LUMBAR HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
OEDEMA (General disorders) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
OESOPHAGITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ORAL BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 3 (3) | 0 (0)
SUPERINFECTION FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TENDON INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
URETERIC INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UTERINE RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN NEOPLASM OF THYMUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CEREBRAL VENOUS SINUS THROMBOSIS (Nervous system disorders) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 1 (1) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 3 (5) | 0 (0)
STATUS MIGRAINOSUS (Nervous system disorders) | 1 (2) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION SUICIDAL (Psychiatric disorders) | 1 (1) | 0 (0)
HALLUCINATION (Psychiatric disorders) | 1 (2) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
TESTICULAR INFARCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
NASAL ULCER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GUTTATE PSORIASIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SHOCK HAEMORRHAGIC (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=680) | Ocrelizumab Safety Follow-up (N=64)
NASOPHARYNGITIS (Infections and infestations) | 210 (449) | 11 (19)
COUGH (Respiratory, thoracic and mediastinal disorders) | 47 (56) | 4 (4)
DIARRHOEA (Gastrointestinal disorders) | 42 (52) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 38 (40) | 0 (0)
FATIGUE (General disorders) | 67 (106) | 0 (0)
PYREXIA (General disorders) | 47 (62) | 0 (0)
INFLUENZA (Infections and infestations) | 92 (137) | 0 (0)
ORAL HERPES (Infections and infestations) | 55 (116) | 0 (0)
SINUSITIS (Infections and infestations) | 36 (58) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 51 (81) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 70 (108) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 294 (569) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 37 (40) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 47 (58) | 0 (0)
HEADACHE (Nervous system disorders) | 154 (320) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 34 (43) | 0 (0)
INSOMNIA (Psychiatric disorders) | 34 (43) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 42 (55) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 57 (74) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-11-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT02861014/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/14/NCT02861014/SAP_001.pdf